CLINICAL TRIAL: NCT01261936
Title: Protocol for the Determination of Menstrual Blood Losses in Women Affected by Congenital Bleeding Disorders
Brief Title: Evaluation of Menses in Congenital Bleeding Disorders
Acronym: MEVA-3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of L'Aquila (Other)
Responsible Party: Napolitano Mariasanta,MD, Ospedale Sna Salvatore-U.O.C. di Medicina Interna ed Ematologia-L'Aquila
Other Study IDs: MEVA-3
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Von Willebrand Disease; Congenital Coagulation Factors Deficiency; Haemophilia Carriers
Keywords: Menorrhagia; Congenital Bleeding Disorders(CBDs); Diagnosis and treatment of menorrhagia in CBDs
MeSH Terms: conditions — von Willebrand Diseases; Menorrhagia; Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vacuum sealed soiled pads and tampons, will be weighted and than opportunely discarghed
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women with a diagnosis of CBD: women in the fertile age, with an ascertained diagnosis of CBD, followed up for heavy periods and needing a specific treatment.

SUMMARY:
Menorrhagia is the term used to define excessive menstrual blood losses, as often based on a subjective judgment of women. Many arbitrary values, expressed in milliliters of blood, have been proposed to define this symptom: 60 on each cycle has also been confirmed in our preliminary study on 87 healthy women. The quantitative determination of menstrual blood losses is nevertheless rarely performed, only in research settings. Although menorrhagia is a quite frequent symptom in healthy women apparently haemostatically competent in the fertile age (20-30%), its incidence becomes very high in women affected by congenital coagulation factors deficiency and (50-62.9%) inherited platelet defects, e.g. Glanzmann's Thromboasthenia (GT); also in von Willebrand Disease the bleeding symptom "menorrhagia" has an high prevalence (60-75%)(8); for GT an incidence of 90% has been reported.

This explains the need for a study focused on the evaluation of menorrhagia in CBDs, addressed to answer to the following, still unsolved questions:

1. Definition of the entity of menstrual blood losses in women affected by CBDs
2. Elaboration of specific treatment schedules for each type of CBD
3. Impact of different specific treatment schedules on kinetic and entity of menstrual losses (how does treatment modify losses?).

DETAILED DESCRIPTION:
The following is a multicentric, observational, cross-over study intended to apply an easy and simple system for the quantitative determination of menstrual losses in women affected by Congenital Bleeding Disorders (CBDs).

The evaluation of menstrual losses represents a scarcely studied field in this specific subset of patients (1), but it is very interesting because of the high incidence of menorrhagia,changeable according to each type of CBDs, but between 60 and 100% in women in the fertile age.

The system adopted for the determination of menstrual losses, called QUEM (QUantitative Evaluation of Menses),is based on the collection of tampons and pads in standard bags which are readily vacuum sealed with a simple device for the whole of woman's period. QUEM has already been validated in preliminary in vitro and ex vivo studies (both in 87 healthy women and in women with CBDs), by comparing it with the gold standard, the Alkaline Haematin Method. A correlation coefficient close to 1 was obtained.

In the current study QUEM will be applied to women in the fertile age (between 18 e 45 years),with an ascertained diagnosis of CBD (FVII, FX, FII deficiencies, Glanzmann and von Willebrand disease, symptomatic Hemophilia A and B carriers), followed up for heavy periods at their reference hemophilia centre and needing a specific treatment will be enrolled in this multicentric study. Also women with apparently normal menses but a severe bleeding disorder will be enrolled. Women with ascertained menorrhagia will be treated with specific replacement therapies, already commonly adopted in clinical practice based on the type of CBD and scheduled to reduce heavy periods.

The study will evaluate 4 consecutive menstrual cycles, the first and the second period without treatment (when possible) and the following two by the administration of the specific treatment.

The bleeding anamnesis (bleeding score) will be performed by applying an international reference method, already validated in von Willebrand Disease type 1 (vWD1) [2] and adopted in an Italian multicentric study on 814 patients affected by different types of VWD [3]. The determination of this score has been considered useful also for other CBDs. This study has already been approved by the IRC of "San Salvatore Hospital"- L'Aquila-Italy. The study is already enrolling, in Italy, women. All the needed materials and equipments will be provided; patients will be carefully informed about the objectives of the study and they will follow a short course illustrating the use and the characteristics of the method proposed (QUEM).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 45 years;
2. Ascertained diagnosis of one of the following inherited bleeding disorders:

   1. Von Willebrand Disease type 1, 2, 3 severe and moderate (VWF:RCo < 30 %),as diagnosed following Italian guidelines [4]
   2. Glanzmann Thromboasthenia
   3. Congenital Coagulation Factor VII, II or X deficiency
   4. A and B Haemophilia Carriers (Factor VIII and IX <25%);
3. Bleeding Severity score > 2
4. Signing the consent form.

Exclusion Criteria:

1. Under continuous anti-hemorrhagic prophylaxis 2. Affected by an active cancer or anti-phospholipid antibodies syndrome 3. History of liver, kidney or endocrine disorders 4. Submucous uterine fibroids, uterine polyps or malignancy 5. Use of oral contraceptives or intrauterine devices in the past three months 6. Treatment with non-steroidal anti-inflammatory drugs

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women affected by CBDs and candidated to receive, as commonly performed in clinical practice a specific substitutive therapy or Desmopressine (rFVIII, rFVIIa, Desmopressine , FVIII concentrates rich in VWF, Activated Prothrombin Complex) will be followed for four consecutive menseses .The number of women enrolled will be between 30 and 50, regardless of parity.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-02; Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Quantitative determination of menstrual blood losses | 1 year
  Quantitative determination of menstrual blood losses in women in the fertile age( between 18 and 45 years) affected by an inherited haemorrhagic disorder diagnosed on the basis of the current International Standard Criteria.This study is preliminary to the evaluation of the efficacy of each

SECONDARY OUTCOMES:
kinetic definition of menses | monthly
  Kinetic definition of menses (hours and days of flow) with and without specific treatment
Influence of treatment on menstrual blood losses | monthly
  To define the influence of substitutive therapies on menstrual losses
treatment schedule evaluation | monthly
  Elaboration of specific treatment schedules for each type of CBD, as evaluated by QUEM

CONTACTS AND LOCATIONS:
Overall Officials: guglielmo mariani, md, Study Director — ospedale "san salvatore"
Locations (3):
- Italy (3):
  - IRCCS "Casa Sollievo della Sofferenza"-Thrombosis and Haemostasis Center, San Giovanni Rotondo, FG
  - Thrombosis and Hemostasis Center-University of L'Aquila, L’Aquila
  - Hematology Department-University of Palermo, Palermo

REFERENCES:
- See also: Diagnosis and treatment of menorrhagia — http://www.asgo.net.au/